CLINICAL TRIAL: NCT05484024
Title: Preoperative Short-course Radiotherapy Followed by Chemotherapy With or Without PD-1 Inhibitor for Locally Advanced Rectal Cancer: a Prospective, Multicenter, Randomized Controlled, Phase II/III Study (STELLAR II Study)
Brief Title: Short-course Radiotherapy Followed by Chemotherapy and PD-1 Inhibitor for Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC22/206-3408
Record Dates: First submitted 2022-07-21; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Rectal Neoplasms Malignant; Radiotherapy
Keywords: rectal cancer; short-course radiotherapy; total neoadjuvant therapy; PD-1 inhibitor
MeSH Terms: conditions — Rectal Neoplasms | interventions — sintilimab; Immune Checkpoint Inhibitors; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTNT group (Experimental): The intervention of iTNT group is Short-course radiotherapy followed by neoadjuvant chemotherapy and PD-1 inhibitor, which consists of a short-course radiotherapy(SCRT, 5 Gy x 5 alone), then after 14 days of radiotherapy completed, four cycles of PD-1 inhibitor and four cycles of CAPOX or six cycles of mFOLFOX will be performed. The regimen of PD-1 inhibitor and CAPOX treatment includes Sintilimab 200 mg IV, day 1，Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle). The regimen of PD-1 inhibitor and mFOLFOX treatment includes Sintilimab 200 mg IV day 1(3 weeks per cycle), Oxaliplatin 85 mg/m2 IV day 1, Leucovorin 400 mg/m2 IV day 1, 5-FU 400 mg/m2 IV bolus on day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) IV continuous infusion(2 weeks per cycle), then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Drug: Sintilimab; Radiation: Short-course radiotherapy; Combination Product: CAPOX/mFOLFOX
- TNT group (Active Comparator): The intervention of TNT group is Short-course radiotherapy followed by neoadjuvant chemotherapy, which consists of a short-course radiotherapy(SCRT, 5 Gy x 5 alone), then after 14 days of radiotherapy completed, four cycles of CAPOX or six cycles of mFOLFOX will be performed. The regimen of CAPOX treatment includes Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle). The regimen of mFOLFOX treatment includes, Oxaliplatin 85 mg/m2 IV day 1, Leucovorin 400 mg/m2 IV day 1, 5-FU 400 mg/m2 IV bolus on day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) IV continuous infusion(2 weeks per cycle), then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Radiation: Short-course radiotherapy; Combination Product: CAPOX/mFOLFOX

INTERVENTIONS:
Drug: Sintilimab — PD-1 inhibitor
  Other Names: Immune checkpoint inhibitor
  Arms: iTNT group
Radiation: Short-course radiotherapy — Pelvic radiation
  Other Names: hypofraction
Combination Product: CAPOX/mFOLFOX — chemotherapy regimen
  Other Names: neoadjuvant chemotherapy

SUMMARY:
This phase II/III trial studies how well neoadjuvant short-course radiotherapy and chemotherapy with or without PD-1 inhibitors works in treating patients with locally advanced rectal adenocarcinoma. Neoadjuvant short-course radiation therapy followed by two-drug regimen chemotherapy, such as CAPOX, were shown to be non-inferior to standard long-course chemoradiotherapy in our previous STELLAR study. Immune checkpoint inhibitors (ICIs) using monoclonal antibodies, such as PD-1 or PD-L1 inhibitor, show promising efficiency and reliable security in some limited sample prospective or retrospective studies. When treating patients with locally advanced rectal cancer, giving sequential neoadjuvant short-course radiotherapy and chemotherapy with PD-1 inhibitor may work better.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven rectal adenocarcinoma;
* Distance between tumour and anal verge≤ 10cm;
* Locally advanced tumour;(8th edition AJCC/UICC staging :cT3-T4N0/cT2-4N+，M0) Cancer Staging must be based on pelvic MRI or Endoscopic ultrasound;
* Eastern Cooperative Oncology Group(ECOG) performance score ≤ 1;
* Mentally and physically fit for chemotherapy; Adequate blood counts: White blood cell count ≥3.5 x 109/L Haemoglobin levels ≥100g/L Platelet count ≥100 x 109/L Creatinine levels ≤1.0× upper normal limit（UNL） Urea nitrogen levels ≤1.0× upper normal limit（UNL） Alanine aminotransferase(ALT) ≤1.5× upper normal limit（UNL） Aspartate aminotransferase(AST) ≤1.5× upper normal limit（UNL） Alkaline phosphatase(ALP) ≤1.5× upper normal limit（UNL） Total bilirubin(TBIL)

  ≤1.5× upper normal limit（UNL）
* No excision of tumor, chemotherapy or other anti-tumor treatment after the diagnosis.
* No previous pelvic radiation history；
* Written informed consent;

Exclusion Criteria:

* Previous treatment with anti-PD-1/L1 and anti-CTLA-4 or other immune experimental drugs.
* Severe autoimmune disease: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (e.g. Wegener's granulomatosis)
* Symptomatic interstitial lung disease or active infectious/non-infectious pneumonia.
* At risk for bowel perforation: active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal cancer or other known risk factors for bowel perforation.
* history of other malignancies, excluding curable non-melanotic skin cancer and cervix carcinoma in situ；
* Active infection, heart failure, heart attack within 6 months, unstable angina or unstable arrhythmia.
* Any condition investigator considered may interfere with the results or place the patient at increased risk of treatment complications, or other uncontrollable disease.
* Pregnancy or breast feeding
* Immunodeficiency disorders including human immunodeficiency virus (HIV), or history of organ transplantation, allogeneic stem cell transplantation
* Active hepatitis B virus (HBV) hepatitis (HBV-DNA ≥ 2000 U/mL), hepatitis C virus (HCV) hepatitis, active tuberculosis infection.
* Oncology vaccination history or any vaccination within 4 weeks prior to the start of treatment.(Note: influenza vaccines are mostly inactivated and therefore allowed, intranasal preparations are usually live attenuated vaccines and therefore not allowed)
* Concomitant other immune agents, chemotherapeutic agents, other drugs in clinical studies, and long term cortisol application

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2022-08-06 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
complete remission | one year
  The rate of pathological complete remission plus clinical complete remission
Disease-free survival rate | three year

SECONDARY OUTCOMES:
Incidence of acute toxicities during radiation, chemotherapy ± immunotherapy | three months
Incidence of surgical complications | 30 days
Overall survival rate | three year
Locoregional recurrence rate | three year
Distance metastasis rate | three year
Radical resection (R0) | one year
Quality of life (QoL) | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using EORTC QLQ-C30 (range 0-100). It evaluates the quality of life from 30 aspects, including appetite, mental status, sleep quality, fatigue, etc. The higher scores mean a better quality of life.
Quality of life (QoL) | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using EORTC QLQ-Cr29 (range 0-100). It evaluates the quality of life from 29 aspects, including defecation function, urine function，pain, sex function, etc. The higher scores mean a better quality of life.
Quality of life (QoL) | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using Wexner score(range 0-20). It evaluates the defecation function. The lower scores mean a better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality
  - National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang Y, Li HY, Wei LC, Li N, Zhang WJ, Lu YF, Deng FY, Xu TZ, Shuai JC, Lei ZF, Meng XY, Qi SN, Song YW, Zhang WW, Jing H, Li G, Liu SX, Wang YJ, Liu Z, Ma HY, Wang NY, Chen B, Wang SL, Li YX, Zhao LN, Tang JQ, Jiang Z, Chen YG, Zhou HT, Hu C, Jin J. Short-course-based TNT with or without PD-1 inhibitor for pMMR locally advanced rectal cancer: Phase 2 results of a randomized trial (STELLAR II). Med. 2025 Nov 14;6(11):100807. doi: 10.1016/j.medj.2025.100807. Epub 2025 Aug 21. PMID 40845854
- [Derived] Zhang W, Tang Y, Wei L, Liu S, Wang W, Chi Y, Wang Y, Kang W, Huang W, Deng F, Li H, Ma H, Jiang L, Ding Z, Feng L, Li Y, Chen Y, Zhou H, Hu C, Jin J. Preoperative short-course radiotherapy followed by chemotherapy and PD-1 inhibitor administration for locally advanced rectal cancer: A study protocol of a randomized phase II/III trial (STELLAR II study). Colorectal Dis. 2024 Sep;26(9):1732-1740. doi: 10.1111/codi.17090. Epub 2024 Jul 17. PMID 39020518